CLINICAL TRIAL: NCT00446342
Title: Phase 1 Multicenter, Dose-Escalation Clinical Study of the Safety and Tolerability of Intravenously Administered SNS-032 Injection, a Novel Cyclin-Dependent Kinase Inhibitor, Administered to Patients With Advanced B-Lymphoid Malignancies
Brief Title: Study of Intravenously Administered SNS-032 in Patients With Advanced B-lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0009
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: B-lymphoid Malignancies; Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma; Multiple Myeloma
Keywords: leukemia; lymphoma; myeloma; non-Hodgkin's; CLL; MCL; MM; Phase 1; hematological malignancy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Multiple Myeloma; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Hematologic Neoplasms | interventions — N-(5-(((5-(1,1-dimethylethyl)-2-oxazolyl)methyl)thio)-2-thiazolyl)-4-piperidinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose-escalation of SNS-032 injection (Experimental): Patients escalated to MTD starting in Cohort 1 of 15 mg/m2 of SNS-032 injection, with 1.5-fold increase each cohort and a maximum loading dose increase of 10 mg/m2. Each dose cohort will have a minimum of 3 patients each with advanced CLL or MM. Dose escalation continues in the absence of Cycle 1 DLT criteria until an MTD is achieved for each disease type to a maximum of 7 cohorts at a high dose of 70 mg/m2. Stage 2 tests at MTD in larger group.
  Interventions: Drug: SNS-032 Injection

INTERVENTIONS:
Drug: SNS-032 Injection — Stage 1: Escalating doses of SNS-032 on days 1, 8 and 15 per 28 day cycle
  Stage 2: Same as stage 1 except SNS-032 administered at the maximum tolerated dose established in stage 1

SUMMARY:
The purpose of this study is to assess the safety and tolerability of escalating doses of SNS-032, given in 3 weekly administrations per cycle and to identify a recommended Phase 2 dose.

DETAILED DESCRIPTION:
Other objectives of this study include measuring pharmacokinetics (how long the drug can be measured in the body) and identifying potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed chronic lymphocytic leukemia (CLL), mantle cell lymphoma (MCL), or multiple myeloma (MM).
* Evidence of relapsed disease
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1

Exclusion Criteria:

* Prior treatment with SNS-032 injection (previously known as BMS-387032)
* Pregnant or breastfeeding
* Unwilling to use an approved, effective means of contraception according to the study site's standards
* Use of therapeutic anticoagulation agents
* Prior allogeneic bone marrow transplantation
* Prior chemotherapy, monoclonal antibodies, investigational agents, or radiation therapy within 21 days before the first dose; nitrosoureas and mitomycin are not permitted for at least 42 days before the first dose.
* Prior pelvic radiation therapy or radiation to > 25% of bone marrow reserve
* Any other medical, psychological, or social condition that would contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures

Please note: There are additional inclusion/exclusion criteria for this study. Please contact the study center for additional information and to determine if the patient meets all study criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of SNS-032 | 1 year

SECONDARY OUTCOMES:
To characterize the pharmacokinetic profile of SNS-032 | 1 year
Identify a recommended Phase 2 dose and schedule of administration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Michelson, MD, Study Director — Sunesis Pharmaceuticals
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Hackensack University Medical Center at the Cancer Center, Hackensack, New Jersey
  - MD Anderson Cancer Center, University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148